CLINICAL TRIAL: NCT03914820
Title: Prophylactic Surgery Plus Hyperthermic Intraperitoneal Chemotherapy (HIPEC CO2) Versus Standard Surgery in Colorectal Carcinoma at High Risk Peritoneal Carcinomatosis. Short and Long-term Outcomes. CHECK STUDY
Brief Title: Prophylactic Surgery Plus HIPEC With CO2 in Patients Affected by Colorectal Carcinoma. CHECK Study.
Acronym: CHECK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-CRC- 7813; 2019-001437-14 (EudraCT Number)
Record Dates: First submitted 2019-04-02; First posted 2019-04-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal cancer; HIPEC CO2; prophylactic surgery; mitomycin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: This is a phase III randomized, multicenter study with two different arm:
  * experimental: prophylactic surgery plus HIPEC CO2 performed with mitomycin
  * comparator: standard surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): ARM A: Prophylactic surgery plus HIPEC CO2 performed with mitomycin
  Interventions: Procedure: HIPEC CO2 surgery; Drug: Mitomycin
- Comparator (Active Comparator): ARM B: Standard surgey without HIPEC CO2 The arm B is with standard surgery without HIPEC CO2
  Interventions: Procedure: Standard surgery

INTERVENTIONS:
Procedure: HIPEC CO2 surgery — Prophylactic surgery plus HIPEC CO2 performed with mitomycin
  Arms: Experimental
Procedure: Standard surgery — Standard surgery without HIPEC CO2
  Arms: Comparator
Drug: Mitomycin — Prophylactic surgery plus HIPEC CO2 performed with mitomycin
  Other Names: HIPEC CO2 surgery with mitomycin
  Arms: Experimental

SUMMARY:
This is a phase III randomized, multicenter study with two different arm:

* experimental: prophylactic surgery plus HIPEC CO2 performed with mitomycin
* comparator: standard surgery Adjuvant treatment after surgery is mandatory except for documented cases of non-eligibility.

Patient will be randomized in a 1:1 ratio. Randomization will be done during surgery if the total resection of tumour will be reached and will use a stratification procedure based on center

DETAILED DESCRIPTION:
This is a phase III randomized, multicenter study with two different arm:

* experimental: prophylactic surgery plus HIPEC CO2 performed with mitomycin
* comparator: standard surgery Adjuvant treatment after surgery is mandatory except for documented cases of non-eligibility.

Patient will be randomized in a 1:1 ratio. Randomization will be done during surgery if the total resection of tumour will be reached and will use a stratification procedure based on center

The HIPEC CO2 regimen will be as reported below:

mitomycin: (total dose of 35 mg/mq, physiologic solution 0.9%) administrated 50% at time 0 from start of HIPEC CO2 treatment (17.5 mg/mq), 25% (8.8 mg/mq) after 30 minutes and the last dose 25% after 60 minutes. Recommended temperature for HIPEC treatment is 41-42 °C for 90 minutes.

Adjuvant treatment consists of a 6 months chemotherapy after surgery. It is possible to choose between Oxaliplatin, Capecitabine (XELOX) or Oxaliplatin, Fluorouracil, Leucovorin (FOLFOX-4) Patients affected by CRC at high risk of developing peritoneal carcinomatosis will be randomized in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented colorectal adenocarcinoma eligible for R0,

   1. Presurgical or intraoperative stage T4a or T4b primary tumour (TNM 8 th)
   2. Urgent presentation: perforation without purulent generalized peritonitis or fecal peritonitis
   3. Peritumoral minimal peritoneal carcinomatosis: limited peritoneal disease in close proximity to the primary tumour, that may be removed en bloc
   4. Ovarian metastases (Krukenberg tumor)
2. Age ≥ 18 and ≤75 years
3. Written informed consent

Exclusion Criteria:

1. Distant metastatic disease (even if limited and completely resected)
2. History of tumour diagnosed in the 3 years before entering the study, except for topical and healed pathologies that do not need further treatment (e.g. non-melanoma skin carcinomas, superficial bladder carcinomas or in situ carcinoma of the breast or cervix).
3. Psychological, family or social conditions which may negatively affect the treatment and follow-up protocol.
4. Poor general conditions (ECOG > 2).
5. Impaired cardiac function (history of congestive heart failure or FE <40%). Clinically significant cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrolment), myocardial infarction (<6 months prior to enrolment), unstable angina, congestive heart failure (New York Heart Association Classification Class > II or serious uncontrolled cardiac Arythmia requiring medication
6. Impaired renal function (creatinine> 1.5 upper limit of normal or creatinine clearance <60 mL / min)
7. Impaired hepatic function (AST, ALT >2.5 upper limit of normal, bilirubin> 1.5 upper limit of normal)
8. Impaired hematopoietic function (leucocytes <4000 / mm3, neutrophils <1500 / mm3, platelets <100000 / mm3)
9. Impaired pulmonary function (presence of COPD or other pulmonary restrictive conditions with FEV1 <50% or DLCO <40% of normal age value).
10. Pregnancy
11. History or presence of other diseases, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of HIPEC or chemotherapy or patient at high risk from treatment complications.
12. Chronic inflammatory bowel disease
13. Patients with acute bowel obstruction
14. Refusal to join the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival (LRFS) | This outcome measure will be assess approximately 3 years after the last patient enrolled
  The primary efficacy endpoint is LRFS defined as the time from randomization to the date of first local relapse, peritoneal carcinomatosis or death for any cause, whichever comes first.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | This outcome measure will be assess approximately 3 years after the last patient enrolled
  Disease Free Survival (DFS) DFS is defined as the time from randomization to the date of first local relapse, distant relapse, peritoneal carcinomatosis or death for any cause, whichever comes first.
  OS is defined as the time from randomization to death for any cause.
Overall Survival (OS) | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  death for any cause
number of post-surgery complication | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  any type of complication
morbidity | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  evaluated during and after surgery, graded according to the NCI-CTAE version 4.03 for AE related to chemotherapy and according to Clavien Dindo for surgery complications
duration of surgery | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  timing of surgery
number of patients performing the adjuvant chemotherapy. | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  patients performing the adjuvant chemotherapy
length of hospitalization | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  length of hospitalization
mortality at 30 and 90 days from surgery | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  mortality at 30 and 90 days from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Pacelli, MD, Principal Investigator — fabio.pacelli@policlinicogemelli.it
Locations (16):
- Italy (16):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - ASP PO Sant'Elia, Caltanissetta
  - AO Santa Croce e Carle, Cuneo
  - ULLS1 1 Dolomiti - Ospedale di Feltre, Feltre
  - Ospedale dell Angelo, Mestre
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Policlinico di Milano, Milan
  - A.O.R.N. A. Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Evangelico Betania, Napoli
  - AOU Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera S. Camillo Forlanini, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Policlinico Universitario Agostino Gemelli Irccs Universita' Cattolica Del Sacro Cuore, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pacelli F, Gerardi C, Rulli E, Abatini C, Rotolo S, Garattini S, Melotti G, Torri V, Galli F, Rulli E, Di Giorgio A; CHECK Investigators. Prophylactic surgery plus hyperthermic intraperitoneal chemotherapy (HIPEC CO2) versus standard surgery in colorectal carcinoma at high risk of peritoneal carcinomatosis: short-term and long-term outcomes from the CHECK study - protocol for a randomised, multicentre, phase 3 trial. BMJ Open. 2022 Aug 1;12(8):e051324. doi: 10.1136/bmjopen-2021-051324. PMID 35914916